CLINICAL TRIAL: NCT04155632
Title: Neurocircuit Strategy to Decrease Cocaine Cue Reactivity
Acronym: COCA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 00091981; 5P50DA046373-04 (NIH)
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- N-acetylcysteine + Theta Burst Stimulation (Experimental)
  Interventions: Drug: N-acetylcysteine; Device: Theta-burst stimulation (TBS)
- N-acetylcysteine + Sham Theta Burst Stimulation (Sham Comparator)
  Interventions: Drug: N-acetylcysteine
- Placebo + Theta Burst Stimulation (Experimental)
  Interventions: Device: Theta-burst stimulation (TBS)
- Placebo + Sham Theta Burst Stimulation (No Intervention)

INTERVENTIONS:
Drug: N-acetylcysteine — N-acetylcysteine (NAC) is a medication that is used to treat paracetamol (acetaminophen) overdose, and to loosen thick mucus in individuals with cystic fibrosis or chronic obstructive pulmonary disease. It has a long-established safety record in adults and children, with FDA approval since 1963. The side effects most commonly noted in people who take NAC by mouth include diarrhea, nausea, vomiting, and headache. These side effects are usually mild and go away even with continued use of NAC by mouth. There is also a risk of a skin reaction, such as flushing, itching, or rash. A meta-analysis of studies evaluating long-term oral treatment with NAC for prevention of chronic bronchitis found that NAC was well tolerated, with generally mild, most commonly gastrointestinal adverse effects that did not require treatment interruption.
  Other Names: NAC
  Arms: N-acetylcysteine + Sham Theta Burst Stimulation; N-acetylcysteine + Theta Burst Stimulation
Device: Theta-burst stimulation (TBS) — Theta-burst stimulation (TBS), a form of repetitive transcranial magnetic stimulation (rTMS), affects brain areas stimulated directly underneath the scalp and brain areas that are functionally connected.
  Arms: N-acetylcysteine + Theta Burst Stimulation; Placebo + Theta Burst Stimulation

SUMMARY:
The overarching goal of this project is to examine the effect of combining theta burst stimulation (TBS) and N-acetylcysteine (NAC) on cocaine craving and brain response to cocaine-related images.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 2. English fluency 4. Meet criteria for cocaine use disorder (CUD), as determined by DSM-V criteria, using the Structured Clinical Interview for DSM-V.

5. Enrolled in an intensive outpatient treatment program (MUSC Center for Drug and Alcohol Programs Intensive Outpatient Program (CDAP-IOP) or currently engaged in treatment for substance related problems.

6. Able to read and understand questionnaires and informed consent 7. Lives within 50 miles of the study site. 8. Is not at elevated risk of seizure (i.e., does not have a history of seizures, is not currently prescribed medications known to lower seizure threshold) 9. Does not have metal objects in the head/neck. 10. Does not have a history of traumatic brain injury, including a head injury that resulted in hospitalization, loss of consciousness for more than 10 minutes, or having ever been informed that they have an epidural, subdural, or subarachnoid hemorrhage.

11. Does not have a history of claustrophobia leading to significant clinical anxiety symptoms.

Exclusion Criteria:

1. Past head injury or primary neurological disorder associated with MRI abnormalities, including dementia, MCI, brain tumors, epilepsy, Parkinson's disease, or demyelinating diseases
2. Any physical or intellectual disability affecting completion of assessments
3. Any contraindication to MRI
4. Current or past psychosis
5. ECT in last 6 months
6. Among females, pregnancy at screening will be exclusionary. Females of child bearing potential must agree to undergo a pregnancy test 72 hours prior to the fMRI scanning session and regularly before and during the medication trial. They must further agree to notify the study physician or PA if they become pregnant during the study.
7. Clinical Institute Withdrawal Assessment (CIWA-Ar) scale will be used to assess alcohol withdrawal. Individuals with CIWA > 8 will be excluded.
8. Individuals with unstable medical illness (e.g., hypertension, diabetes, myocardial infarction)
9. Has current suicidal ideation or homicidal ideation.
10. Has the need for maintenance or acute treatment with any psychoactive medication including anti-seizure medications and medications for ADHD
11. Suffers from chronic migraines
12. Any physical or intellectual disability affecting completion of assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: All Validations Passed Badran, PhD, Principal Investigator — Medical University of SC
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only 32 were randomized and started treatment.
Groups:
- Active Theta Burst Stimulation: Two trains of 120-second active cTBS consisted of 3-pulse bursts delivered at 5 Hz.
- Sham Theta Burst Stimulation: Two trains of 120-second sham cTBS consisted of 3-pulse bursts delivered at 5 Hz.
Period: Overall Study
Arm/Group | Active Theta Burst Stimulation | Sham Theta Burst Stimulation
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Theta Burst Stimulation | Sham Theta Burst Stimulation | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: year] | 48.3 (10.5) | 53.8 (10.9) | 51.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 11 | 14 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 11 | 19
  White | 7 | 4 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Cocaine Craving Rating [Mean (Standard Deviation); unit: score on a scale] — Self-reported craving measured using a Numerical Rating Scale (NRS) from 1 to 10, where 1 = no craving and 10 = extreme craving. Higher scores indicate greater craving.
  score on a scale | 4.39 (2.04) | 4.45 (1.98) | 4.42 (1.98)
Profile of Mood States (POMS) [Mean (Standard Deviation); unit: POMS score] — Profile of Mood States (POMS) total score, ranging from 0 to 200. Higher scores indicate greater mood disturbance. Subscales include tension, depression, anger, vigor, fatigue, and confusion
  POMS score | 23.50 (34.86) | 18.75 (30.95) | 21.13 (32.52)
OFC brain activity [Mean (Standard Deviation); unit: Percent BOLD signal change] — Measured using fMRI during cocaine cue reactivity task. Percent signal change in orbitofrontal cortex (OFC) during cocaine vs. neutral image blocks.
  Percent BOLD signal change | 0.0049 (0.0096) | -0.0012 (0.0102) | 0.0018 (0.0102)

OUTCOME MEASURES:

1. Primary Outcome: Change in Orbitofrontal Cortex (OFC) BOLD Signal During Cocaine Cue Reactivity Task (Pre- vs. Post-TBS)
Description: Measured using fMRI during cocaine cue reactivity task. Percent BOLD signal change in OFC from baseline (Visit 2) to post-TBS (Visit 3). Measured using functional MRI during a cocaine cue reactivity task. The outcome reflects the change in raw BOLD signal in the orbitofrontal cortex (OFC) between baseline and post-TBS sessions. Signal change was calculated by comparing activation during cocaine-related image blocks versus neutral image blocks. Values are reported as raw BOLD signal units (not percentages).
Time Frame: From baseline to immediately post-TBS
Measure: Mean (Standard Deviation); unit: BOLD signal
Arm/Group | Active Theta Burst Stimulation | Sham Theta Burst Stimulation
Number analyzed (Participants) | 16 | 16
BOLD signal | -0.0026 (0.0080) | 0.0007 (0.0105)

2. Primary Outcome: Change in POMS Score From Baseline to Post-TBS"
Description: Total POMS score measured before and after TBS. Higher scores indicate worse mood.
Time Frame: From baseline to immediately post-TBS
Measure: Mean (Standard Deviation); unit: POMS score
Arm/Group | Active Theta Burst Stimulation | Sham Theta Burst Stimulation
Number analyzed (Participants) | 16 | 16
POMS score | 5.53 (27.58) | 14.63 (23.32)

3. Primary Outcome: Change in Cocaine Craving Rating From Baseline to Post-TBS
Description: Self-reported craving measured using NRS (1-10) before and after TBS. Higher scores indicate greater craving.
Time Frame: From baseline to immediately post-TBS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Theta Burst Stimulation | Sham Theta Burst Stimulation
Number analyzed (Participants) | 16 | 16
score on a scale | 3.31 (2.32) | 3.99 (2.43)

ADVERSE EVENTS:
Time Frame: From baseline (Visit 2) through 3 weeks post-TBS (Visit 3), including follow-up calls at 1 day, 1 week, 2 weeks, and 3 weeks.
Arm/Group | Active Theta Burst Stimulation | Sham Theta Burst Stimulation
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

LIMITATIONS AND CAVEATS:
We only investigate a single session of cTBS in participants with CUD. Repeated cTBS sessions may produce long-lasting changes in craving and relapse prevention, which should be explored in future research.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT04155632/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT04155632/ICF_001.pdf